CLINICAL TRIAL: NCT04337190
Title: Impact of Previous Treatment With Angiotensin II Receptor Blockers in Patients With SARS-Cov2 Infection Admitted to the Intensive Care Unit on Survival and Severity of the Disease (COVID-ARA2)
Brief Title: Impact of Angiotensin II Receptor Blockers Treatment in Patients With COVID 19 (COVID-ARA2)
Acronym: COVID-ARA2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVID-ARA2
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: COVID; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for measurement of ACE 2 level and ACE 2 activity (ratio Angiotensin(1-7)/Angiotensin(1-10))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sampling — blood sampling at the day of admission, day 3 and day 7

SUMMARY:
The actual pandemic infection related to SARS-CoV2 results in viral pneumonitis (COVID-19), that may, in the more severe cases, lead the patients to the intensive care unit (ICU). The more frequent presentation is acute respiratory distress syndrome (ARDS).

To penetrate cells, SARS-CoV2 uses Angioconvertase type 2 (ACE2) as a cellular entry receptor.

ACE2 belong to the renin-angiotensin-aldosteron system (SRAA), and ACE2 levels are directly modified when SRAA inhibitors are administred to patients, and ACE2 level increases particularely with Angiotensin II Receptor blockers (ARA2) use.

The aim of our study is to determine ACE2 level and activity in patients with SARSCoV2 infection admitted to the intensive care unit (ICU).

COVID ARA2 is a propsective cohort of patient with blood sampling at the day of admission, day 3 and day 7.

DETAILED DESCRIPTION:
The actual pandemic infection related to SARS-CoV2 results in viral pneumonitis (COVID-19), that may, in the more severe cases, lead the patients to the intensive care unit (ICU). The more frequent presentation is acute respiratory distress syndrome (ARDS).

To penetrate cells, SARS-CoV2 uses Angioconvertase type 2 (ACE2) as a cellular entry receptor.

ACE2 belong to the renin-angiotensin-aldosteron system (SRAA), and ACE2 levels are directly modified when SRAA inhibitors are administred to patients, and ACE2 level increases particularely with Angiotensin II Receptor Blockers (ARA2) use.

The aim of our study is to determine ACE2 level and activity in patients with SARSCoV2 infection admitted to the intensive care unit (ICU).

COVID ARA2 is a propsective cohort of patient with blood sampling at the day of admission, day 3 and day 7.

ELIGIBILITY:
Inclusion Criteria:

* admission to the intensive care unit,
* with a proven COVID infection, responsible for acute respiratory failure
* agree with participation to the study.

Exclusion Criteria:

* aged under 18
* under legal protection
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants :
  * will be admitted to the ICU for respiratory failure in a context of proven COVID.
  * will be, or not, treated for chronic hypertension,
  * will need, or not, mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-10-06 (Estimated); Study Completion 2020-12-06 (Estimated)

PRIMARY OUTCOMES:
ACE2 level change over time | at the day of admission, day 3 and day 7
  ELISA test (Higher the ACE2 level, higher the virus penetrate cells)

SECONDARY OUTCOMES:
ACE2 activity over time | at the day of admission, day 3 and day 7
  Ratio angiotensin (1-7)/angiotensin(1/10) (Higher Ratio angiotensin (1-7)/angiotensin(1/10), higher is ACE2 activity)
Mortality at day 28 | day 28
  Mortality at day 28
ARDS severity | from the day of admission to day 7
  PaO2/FiO2 ratio (ARDS is severe when <100, moderate when between 100 and 200, mild when >200)
Duration of mechanical ventilation | from the day of admission to day 28
  Day under mechanical ventilation
Need for prone positionning | from the day of admission to day 28
  Need for prone positionning
Need for extracorporeal membran oxygenation | from the day of admission to day 28
  Need for extracorporeal membran oxygenation
Use of paralytic agents | from the day of admission to day 28
  Need for use of paralytic agents
Need for renal replacement therapy | from the day of admission to day 28
  Need for renal replacement therapy
Need for vasoactive drugs (norepinephrine, dobutamine,epinephrine) | from the day of admission to day 28
  Need for vasoactive drugs
Sequential Organ Failure Assessment (SOFA) score | from the day of admission to day 7
  The SOFA score evaluates the severity of patients through 6 items: respiration (PaO2/FiO2 ratio); coagulation (platelets count); liver (bilirubin); Cardiovascular (hypotension); Central nervous system (coma glasgow score) and Renal (creatinine serum level). Score ranges from 0 to 24, a higher score indicates higher severity and probability of death
Number of session(s) of prone positionning | from the day of admission to day 28
  Number of session(s) of prone positionning
Duration of extracorporeal membran oxygenation treatment | from the day of admission to day 28
  Duration of extracorporeal membran oxygenation treatment
Type of vasoactive drugs | from the day of admission to day 28
  Several vasoactive agents may be used: norepinephrine, dobutamine, epinephrine, vasopressin analogues...
Duration of vasoactive treatment | from the day of admission to day 28
  Duration of vasoactive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Asfar, MD, PhD, Principal Investigator — CHU Angers, service de médecine intensive réanimation
Locations (1):
- University Hospital Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No